CLINICAL TRIAL: NCT06968988
Title: Phase I Study With Expansion Cohort of Zanzalintinib in Combination With Ipilimumab and Nivolumab in Patients With Metastatic Soft Tissue Sarcoma
Brief Title: Zanzalintinib in Combination With Ipilimumab and Nivolumab in Patients With Metastatic Soft Tissue Sarcoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202507090
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Soft-tissue Sarcoma
Keywords: Soft Tissue Sarcoma; Zanzalintinib; Immunotherapy; Nivolumab; Ipilimumab
MeSH Terms: conditions — Sarcoma | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dose Escalation Dose Level 1 (starting dose): Zanzalintinib + Nivolumab + Ipilimumab (Experimental): Zanzalintinib 40 mg by mouth once per day is self administered daily, and nivolumab 3 mg/kg intravenously and ipilimumab 1 mg/kg intravenously are administered intravenously every 3 weeks for a total of 4 doses. After completion of the first 4 cycles, ipilimumab is discontinued while nivolumab 480 mg intravenously is continued every 4 weeks in combination with daily zanzalintinib.
  Interventions: Drug: Zanzalintinib; Drug: Ipilimumab; Drug: Nivolumab
- Dose Escalation Dose Level 2: Zanzalintinib + Nivolumab + Ipilimumab (Experimental): Zanzalintinib 60 mg by mouth once per day is self administered daily, and nivolumab 3 mg/kg intravenously and ipilimumab 1 mg/kg intravenously are administered intravenously every 3 weeks for a total of 4 doses. After completion of the first 4 cycles, ipilimumab is discontinued while nivolumab 480 mg intravenously is continued every 4 weeks in combination with daily zanzalintinib.
  Interventions: Drug: Zanzalintinib; Drug: Ipilimumab; Drug: Nivolumab
- Dose Escalation Dose Level -1: Zanzalintinib + Nivolumab + Ipilimumab (Experimental): Zanzalintinib 20 mg by mouth once per day is self administered daily, and nivolumab 3 mg/kg intravenously and ipilimumab 1 mg/kg intravenously are administered intravenously every 3 weeks for a total of 4 doses. After completion of the first 4 cycles, ipilimumab is discontinued while nivolumab 480 mg intravenously is continued every 4 weeks in combination with daily zanzalintinib.
  Interventions: Drug: Zanzalintinib; Drug: Ipilimumab; Drug: Nivolumab
- Expansion: Zanzalintinib + Nivolumab + Ipilimumab (Experimental): Zanzalintinib dose determined in Dose Escalation by mouth once per day is self administered daily, and nivolumab 3 mg/kg intravenously and ipilimumab 1 mg/kg intravenously are administered intravenously every 3 weeks for a total of 4 doses. After completion of the first 4 cycles, ipilimumab is discontinued while nivolumab 480 mg intravenously is continued every 4 weeks in combination with daily zanzalintinib.
  Interventions: Drug: Zanzalintinib; Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Zanzalintinib — Zanzalintinib will be supplied by Exelixis, Inc.
  Other Names: XL092
Drug: Ipilimumab — Ipilimumab will be commercially sourced.
  Other Names: Yervoy
Drug: Nivolumab — Nivolumab will be commercially sourced.
  Other Names: Opdivo

SUMMARY:
The investigators hypothesize that zanzalintinib in combination with ipilimumab and nivolumab will be well tolerated and serve as a potential therapeutic strategy in metastatic soft tissue sarcoma (mSTS) including myxofibrosarcoma, undifferentiated pleomorphic sarcoma, dedifferentiated liposarcoma, cutaneous angiosarcoma, and undifferentiated sarcoma histologies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed soft tissue sarcoma that is metastatic or unresectable.
* Must have received at least one but no more than 3 lines of therapy in the metastatic setting, with progression on last line of therapy. Neoadjuvant or adjuvant therapy completed more than one year prior does not count towards as a line of therapy in the metastatic. Individuals with alveolar soft part sarcoma may enroll without being refractory to at least one line of therapy.
* Measurable disease per RECIST 1.1.
* At least 18 years of age.
* ECOG performance status ≤ 1.
* Adequate bone marrow and organ function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1.5 K/cumm without granulocyte colony-stimulating factor support within 2 weeks prior to screening laboratory collection
  * Platelets ≥ 100 K/cumm without transfusion within 2 weeks prior to screening laboratory collection
  * Hemoglobin ≥ 9.0 g/dL without transfusion within 2 weeks prior to screening laboratory collection
  * INR ≤ 1.5 and aPTT ≤ 1.2 x IULN. For subjects on Factor Xa inhibitors, criteria does not apply.
  * Total bilirubin ≤ 1.5 x IULN (for subjects with Gilbert's disease ≤ 3 x IULN)
  * AST(SGOT), ALT(SGPT), and alkaline phosphatase (ALP) ≤ 3.0 x IULN. For subjects with documented bone metastasis, ALP ≤ 5.0 x IULN.
  * Serum albumin ≥ 2.8 g/dL.
  * Calculated creatinine clearance ≥ 40 mL/min by Cockcroft-Gault.
  * UPCR ≤ 1 mg/mg (≤ 113.2 mg/mmol) creatinine.
* Recovery to baseline or ≤ grade 1 from AEs, including immune-related AEs related to any prior treatments, unless AEs are clinically nonsignificant and/or stable on supportive therapy (e.g., physiological replacement of corticosteroid). Low-grade or controlled toxicities such as alopecia, ≤ grade 2 hypomagnesemia, ≤ grade 2 neuropathy are permitted.
* Sexually active fertile subjects and their partners must agree to use highly effective method of contraception during the course of the study and for the following durations after the last dose of treatment (whichever is later). An additional contraceptive method, such as a barrier method (eg, condom), is required. In addition, men must agree not to donate sperm and women must agree not to donate eggs (ova, oocyte) for the purpose of reproduction during these same periods:

  * 186 days after last dose of zanzalintinib (for women) or 96 days after last dose of zanzalintinib (for men).
  * 5 months after the last dose of nivolumab or 3 months after the last dose of ipilimumab.
* Female subjects of childbearing potential must not be pregnant at screening. Female subjects are considered to be of childbearing potential unless one of the following criteria is met: permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal status (defined as 12 months of amenorrhea in a woman > 45 years-of-age in the absence of other biological or physiological causes. In addition, females < 55 years-of-age must have a serum follicle stimulating hormone [FSH] level > 40 mIU/mL to confirm menopause). Note: Documentation may include review of medical records, medical examination, or medical history interview by study site staff.
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Translocation-driven sarcoma except for ASPS.
* Prior treatment with zanzalintinib, cabozantinib, PD-1 inhibitor (eg, cemiplimab, nivolumab, pembrolizumab), PD-L1 inhibitor (eg, atezolizumab, avelumab, durvalumab), or CTLA-4 inhibitor (eg, ipilimumab).
* Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before first dose of study treatment.
* Receipt of any type of cytotoxic, biologic, or other systemic anticancer therapy (including investigational) within 4 weeks before first dose of study treatment.
* Radiation therapy for bone metastasis within 2 weeks before first dose of study treatment; any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before first dose of study treatment. Note: Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of enrollment. Note: Base of skull lesions without definitive evidence of dural or brain parenchymal involvement are allowed.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to zanzalintinib, ipilimumab, nivolumab, or other agents used in the study.
* Concomitant anticoagulation with warfarin or other vitamin-K antagonists, direct thrombin inhibitors, or antiplatelet agents (e.g. clopidogrel). Allowed anticoagulants are the following:

  * Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
  * Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen. Note: subjects must have discontinued oral anticoagulants within 3 days or 5 half-lives prior to first dose of study treatment, whichever is longer.
* Any complementary medications (e.g. herbal supplements or traditional Chinese medicines) to treat the disease under study within 2 weeks before first dose of study treatment.
* Uncontrolled, significant intercurrent or recent illness including, but not limited to:

  * Unstable or deteriorating cardiovascular disorders:

    * Congestive heart failure NYHA Class 3 or 4, or Class 2 or higher unstable angina pectoris, new-onset angina, serious cardiac arrhythmias (e.g. ventricular flutter, ventricular fibrillation, Torsades de pointes).
    * Uncontrolled hypertension defined as sustained blood pressure > 140 mmHg systolic or > 90 mmHg diastolic despite optimal antihypertensive treatment.
    * Stroke (including transient ischemic attack), myocardial infarction, or other clinically significant arterial thrombotic and/or ischemic event within 6 months before first dose of study treatment.
    * Pulmonary embolism or deep vein thrombosis or prior clinically significant venous events within 3 months before first dose of study treatment. Note: Subjects with a diagnosis of DVT within 6 months are allowed if asymptomatic and stable at screening and are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen. Note: Subjects who don't require prior anticoagulation therapy may be eligible but must be discussed and approved by the PI.
    * Prior history of myocarditis.
  * Gastrointestinal disorders, including those associated with a high risk of perforation or fistula formation:

    * Tumors invading the GI tract from external viscera
    * Active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, or acute pancreatitis
    * Acute obstruction of the bowel, gastric outlet, or pancreatic or biliary duct within 6 months before first dose unless cause of obstruction is definitively managed and subject is asymptomatic.
    * Abdominal fistula, gastrointestinal perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose. Note: complete healing of an intra-abdominal abscess must be confirmed before first dose of study treatment.
    * Known gastric or esophageal varices.
    * Ascites, pleural effusion, or pericardial fluid requiring drainage in last 4 weeks.
* Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 mL) of red blood, or other history of significant bleeding (e.g. pulmonary hemorrhage) within 12 weeks before first dose of study treatment.
* Symptomatic cavitating pulmonary lesion(s) or endobronchial disease (asymptomatic or radiated lesions allowed).
* Lesions invading major blood vessel including, but not limited to, inferior vena cava, pulmonary artery, or aorta. Note: subjects with intravascular tumor extension (e.g. tumor thrombus in renal vein on inferior vena cava) may be eligible following PI approval.
* Other clinically significant disorders that would preclude safe study participation, in the opinion of the investigator. Specific conditions are noted below:

  * Active infection requiring systemic treatment. Note: prophylactic antimicrobial treatments (antibiotics, antimycotics, antivirals) are allowed.
  * Known infection with acute or chronic hepatitis B or C, known HIV or AIDS-related illness except for subjects meeting all of the following criteria:

    * On stable anti-retroviral therapy
    * CD4+ T cell count ≥ 200/μL
    * Undetectable viral load. Note: HIV testing will be performed at screening if and as required by local regulation. Note: to be eligible, participants taking CYP inhibitors (e.g. zidovudine, ritonavir, cobicistat, didanosine) orCYP3 inducers (efavirenz) must change to a different regimen not including these drugs 7 days prior to initiation of study treatment. Anti-retroviral therapies must have been received for at least 4 weeks prior to the first dose. Note: CD4+ T cell counts and viral load are monitored per standard of care by the local health provider.
  * Serious non-healing wound/ulcer/bone fracture. Note: non-healing wounds or ulcers are permitted if due to tumor-associated skin lesions.
  * Malabsorption syndrome.
  * Pharmacologically uncompensated, symptomatic hypothyroidism.
  * Moderate to severe hepatic impairment (Child-Pugh B or C).
  * Requirement for hemodialysis or peritoneal dialysis.
  * History of solid organ or allogeneic stem cell transplant.
* Major surgery (e.g. GI surgery, removal or biopsy of brain metastasis) within 8 weeks prior to first dose of study treatment. Prior laparoscopic surgeries (e.g. nephrectomy) within 4 weeks prior to first dose of study treatment. Minor surgery (e.g. simple excision, tooth extraction) within 5 days before first dose of study treatment. Complete wound healing from major or minor surgery must have occurred at least prior to first dose of study treatment. Note: fresh tumor biopsies should be performed at least 5 days before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgical procedures, including biopsies, are not eligible.
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 480 ms within 14 days per ECG before first dose of study treatment. Note: triplicate ECG evaluations will be performed and the average of these 3 consecutive results for QTcF will be used to determine eligibility.
* History of psychiatric illness likely to interfere with ability to comply with protocol requirements or give informed consent.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test within 14 days of study entry.
* Inability to swallow tablets or ingest a suspension either orally or by a NG or PEG tube.
* Another malignancy that requires active therapy and in the opinion of the Investigator would interfere with monitoring of radiologic assessments of response to study treatment, within 2 years before first dose of study treatment, except for superficial skin cancers, or localized, low-grade tumors deemed cured and not treated with systemic therapy
* Any active, known, or suspected autoimmune disease. Note: subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger, or permitted to enroll.
* Known positive test for tuberculosis infection if supported by clinical or radiographic evidence of disease.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (eg, bronchiolitis obliterans), drug induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computerized tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Free thyroxine (FT4) outside the laboratory normal reference range. Asymptomatic subjects with FT4 abnormalities can be eligible after Principal Investigator approval.
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy (> 10 mg daily prednisone equivalent) or any other form of immunosuppressive therapy within 2 weeks prior to first dose of study treatment. Inhaled, intranasal, intraarticular, and topical corticosteroids and mineralocorticoids are allowed. Note: Adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease. Transient short-term use of higher doses of systemic corticosteroids for allergic conditions (eg, contrast allergy) is also allowed.
* Administration of a live, attenuated vaccine within 30 days before first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2026-08-12 (Estimated); Study Completion 2031-07-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of dose-limiting toxicities (DLTs) | Through day 42
  DLTs are defined in the protocol.

SECONDARY OUTCOMES:
Frequency and grades of treatment-emergent adverse events (TEAEs) | From start of treatment through 100 days after completion of treatment (estimated to be 24 months and 100 days)
  Graded per CTCAE v5.0.
Rate of treatment discontinuation due to treatment-emergent adverse events (TEAEs) | From start of treatment through completion of treatment (estimated to be 24 months)
Objective response rate (ORR) per RECIST 1.1 criteria | Through completion of treatment (estimated to be 24 months)
  * Objective response (OR) is defined as number of participants with complete response (CR) or partial response (PR).
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Clinical benefit rate (CBR) per RECIST 1.1 criteria | Through completion of treatment (estimated to be 24 months)
  * Clinical benefit is defined complete response (CR), partial response (PR) or stable disease (SD) for 6 weeks.
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Duration of response (DoR) | Through completion of follow-up (estimated to be 60 months)
  * DOR is time from treatment initiation to disease progression or death as a first event for patients who achieve a complete response (CR) or partial response (PR).
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

CONTACTS AND LOCATIONS:
Overall Officials: Mia Weiss, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (IPD) underlying the results reported in this article, including text, tables, figures, and appendices, will be made available. In addition, the study protocol, statistical analysis plan, and informed consent form will be available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be accessible beginning 6 months and ending 36 months following publication of the article
Access Criteria: Access will be granted to researchers who provide a methodologically sound proposal that aligns with the aims outlined in the approved proposal. The data will be shared specifically for analyses that achieve these aims. Researchers interested in accessing the data should submit a proposal to bvantine@wustl.edu. Following approval of the proposal and completion of a data access agreement, the requested data will be provided.
URL: http://siteman.wustl.edu

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu